CLINICAL TRIAL: NCT02125734
Title: A Randomized, Multicenter, Open-label, Cross-over Study to Assess Lung Function and Patient Preference After a 4 Week Treatment Each With QVA149 vs. Tiotropium in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD) and Moderate to Severe Airflow Limitation Who Are on a Tiotropium Therapy (FAVOR Study)
Brief Title: Lung Function and Patient Preference With QVA149 vs. Tiotropium in COPD Patients
Acronym: FAVOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CQVA149ADE04; 2013-004223-37 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Experimental): QVA149 from day 1 to day 28 and tiotropium from day 29 to day 56
  Interventions: Drug: QVA149; Drug: Tiotropium
- Treatment sequence 2 (Experimental): Tiotropium from day 1 to day 28 and QVA149 from day 29 to day 56
  Interventions: Drug: QVA149; Drug: Tiotropium

INTERVENTIONS:
Drug: QVA149 — QVA149 capsules 110/50 µg for inhalation via Concep-1-inhaler device, taken once a day
  Other Names: indacaterol maleate/glycoporromium bromide
Drug: Tiotropium — Tiotropium 18 µg capsules for inhalation via HandiHaler device taken once a day

SUMMARY:
The study is a multicenter, randomized, 2-period, open-label, two arm, cross-over study to show the superior effect of a 4 week treatment each with QVA149 versus tiotropium on lung function. Similarly, this study aims to evaluate patient preference after experiencing both treatment regimens in patients with a clinical diagnosis of COPD (GOLD 2013) and a moderate to severe airflow limitation who are symptomatic (defined as CAT score of at least 10) at screening despite being treated with tiotropium

ELIGIBILITY:
Inclusion Criteria:

* signed an Informed Consent Form
* stable COPD according to current guidelines (GOLD 2013)
* airflow limitation indicated by a post-bronchodilator FEV1/FVC ratio of <0.70 and a post-bronchodilator FEV1 of ≥30% and <80% of predicted normal values at Visit 2.
* current or ex-smokers who have a smoking history of at least 10 pack years
* Patients on stable tiotropium (18 µg/d) monotherapy for at least 8 weeks before Visit 1
* Symptomatic patients defined as patients with CAT score ≥ 10 at Visit 1 (Screening).

Exclusion Criteria:

* Pregnant or breast feeding mothers
* Patients with conditions contraindicated for treatment
* Patients with a history of clinically significant diseases
* Patients who have a clinically significant renal disease
* Patients with myocardial infarctions less than 6 months prior to study entry
* Patients with recent (less than 1 year) history of NYHA Class III/IV left ventricular failure.
* Patients with narrow-angle glaucoma, symptomatic prostatic hyperplasia or bladder-neck obstruction or urinary retention
* Patients with a history of malignancy of any organ system
* Patients who have had a COPD exacerbation that required treatment with antibiotics, and/or systemic steroids (oral or intravenous) and/or hospitalization in the 6 weeks prior to Screening
* Patients who have had a respiratory tract infection within 6 weeks prior to Screening
* Patients with any history of asthma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Germany (16):
  - Novartis Investigative Site, Ibbenbüren, Rhineland-Palatinate
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Garmisch-Partenkirchen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Sonneberg
  - Novartis Investigative Site, Warendorf

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 40 | 48
Completed | 40 | 48
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 40 | 48
Completed | 40 | 47
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Total
Number analyzed (Participants) | 40 | 48 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.83) | 66.0 (9.31) | 65 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 25 | 32 | 57

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) at 1 h Post-inhalation
Description: Forced Expiratory Volume in one second (FEV1) will be calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
Time Frame: week 4
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 87 | 88
Liters | 1.676 (0.5709) [1.635 to 1.716] | 1.595 (0.6000) [1.555 to 1.634]
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Net) = 0.081, 95% CI 2-sided [0.031 to 0.130]

2. Secondary Outcome: Patient Preference After Experiencing Both Treatments Was Assessed at the End of Treatment Period 2 With a Patient Preference Questionnaire.
Description: Patient preference after experiencing both treatments. The patient's preference questionnaire was a two-choice question (preference for QVA149 OR Tiotropium.
Time Frame: 8 weeks
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. Three patients were missing data for the patient preference analysis.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 85 | 85
Participants | 59 | 26

3. Secondary Outcome: Investigator Preference Per Patient After Experiencing Both Treatments for Future Suggestions.
Description: The investigator preference for future treatment suggestion after experiencing both treatments was assessed at the end of treatment period 2 with the Investigator Preference Questionnaire
Time Frame: 8 weeks
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. One patient with missing data for this analysis.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 87 | 87
Participants | 71 | 16

ADVERSE EVENTS:
Groups:
- QVA149: QVA149
- Tiotropium: Tiotropium
Arm/Group | QVA149 | Tiotropium
Serious Adverse Events (participants affected / at risk) | 1/88 | 0/88
Other Adverse Events (participants affected / at risk) | 28/88 | 21/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=88) | Tiotropium (N=88)
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=88) | Tiotropium (N=88)
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Escherichia test positive (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 2
Hypotonia (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety